CLINICAL TRIAL: NCT00594282
Title: Use of a Radiolucent Pad to Reduce Mammography Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Kim K. Engelman, PhD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 9673; POP053504
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Enhanced Mammography (EM) - Women who are randomized to the Enhanced Mammography (EM) condition will receive a mammogram in which a MammoPad radiolucent breast plate cushion is used.
  Interventions: Device: Radiolucent cushion
- 2 (No Intervention): Routine Mammography (RM) - Women who are randomized to the Routine Mammography (RM) condition will obtain a routine, un-altered mammogram during which typical exam protocol will be followed and no radiolucent cushion is used.

INTERVENTIONS:
Device: Radiolucent cushion — MammoPad radiolucent breast plate cushion used during mammogram
  Arms: 1

SUMMARY:
The objective of this study is to assess whether use of a mammography breast plate cushion will significantly decrease the level of discomfort experienced by African American women during routine screening mammograms. The primary hypothesis is that use of the breast plate cushion will result in less mammography-related discomfort. The secondary hypotheses are that women who anticipate high levels of discomfort will experience greater reductions in discomfort when a breast plate cushion is used and participants who received mammograms using a breast plate cushion will have greater intentions to return for a routine mammogram than the control group.

DETAILED DESCRIPTION:
Despite improvements over the past decade, routine mammography screening rates among African American women remain suboptimal. This is especially troubling in light of the fact that African American women have higher breast cancer mortality rates than White and Hispanic women. Multiple studies have revealed that women experience varying levels of pain during mammography, however, African American women report higher levels of mammography-related pain than their White counterparts. In fact, the fear of pain associated with mammography is so prominent that it prevents some women from undergoing routine screenings or follow-ups. Since pain is a major barrier for many African American women in the screening process, studies to assess methods to reduce mammography-related pain are imperative. An FDA-approved radiolucent breast plate cushion has been developed for use during mammography to increase comfort during the exam. The purpose of this study is to evaluate whether use of this radiolucent cushion will decrease the level of pain experienced by African American women undergoing routine screening mammography, positively impact routine mammography screening intentions, and result in greater mammography satisfaction among African American women. 304 women scheduled for mammograms at three community metropolitan mammography facilities participated in this study. One-half of the women were randomized to an Enhanced Mammography (EM) condition in which a radiolucent cushion was used during mammograms. The other half were randomized to a Routine Mammography (RM) condition during which typical exam protocol is followed and no radiolucent cushion was used. Pre- and post-exam surveys assessed anticipated and experienced exam-related pain and discomfort, intentions to return for a future routine mammogram, and general visit satisfaction. A follow-up telephone interview will be conducted with study participants to determine whether they received a follow-up routine screening mammogram 12 to 18 months after they were enrolled in the study (at the time of their last routine screening mammogram) and where they received their mammogram (e.g. did they return to the same facility). If they did not obtain an on-time routine screening mammogram barriers were assessed. The RM and EM groups will be compared for differences.

ELIGIBILITY:
Inclusion Criteria:

* African American women
* 40 years of age or older who presented for a routine screening mammogram

Exclusion Criteria:

* Males
* race other than African American
* younger than 40 years of age

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
A Pre-Mammography Survey and Post-Mammography Survey to assess anticipated and actual discomfort

SECONDARY OUTCOMES:
Pre-Mammography Survey, Post-Mammography Survey to assess barriers

CONTACTS AND LOCATIONS:
Overall Officials: Kim K. Engelman, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States